CLINICAL TRIAL: NCT04297657
Title: THE EFFECT OF BETTER MODEL COUNSELLING WITH MODEL OVER SEXUAL PROBLEMS OF WOMEN WITH BREAST CANCER
Brief Title: Using BETTER Model Sexual Problems in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Zeynep Olcer, PhD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Istanbul University
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Sexuality; Breast Cancer
Keywords: breast cancer; sexuality; better model; nursing care
MeSH Terms: conditions — Sexuality; Breast Neoplasms | interventions — Counseling; Educational Status

STUDY DESIGN:
Intervention Model Description: pre evaluation-final evaluation, control group work
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Counselling
- control group (No Intervention)

INTERVENTIONS:
Other: Counselling — o An appointment was made with the women in the experimental group at a time when they were available and a suitable environment was arranged in the hospital. The counselling programme of the experimental group was conducted in four sessions one week apart. In addition, each woman in the experimental group was given a counselling booklet and compact disc. The interviews lasted between 15- 45 minutes. The topics of interest among women were noted in the interviews and after the information on the subject was received, feedback was given to the relevant woman through a phone call.
  Other Names: education
  Arms: intervention group

SUMMARY:
Breast cancer and its treatments such as mastectomy, chemotherapy, radiotherapy, hormonal therapy cause many side effects such as scar, problems with body perception and sexual problems. Sexual concerns lead to significant emotional distress, including sadness/depression, issues related to personal appearance, stigma, and negative impacts on personal relationships, intimacy and sexuality all of which reduce the quality of life. This experimental type of research is conducted within the framework of the BETTER model to evaluate the impact of counselling programme on sexuality issues that patients with breast cancer experience.

DETAILED DESCRIPTION:
Methods: The sampling consists of 60 female participants who volunteered to participate in the study. Face to face interviews are held with the female participants based on the Information Forms and Female Sexual Function Index (FSFI)", "EORTC QLQ-BR23 Quality of Life Questionnaire", "Center for Epidemiologic Studies Depression Scale (CES-D)", "Body Cathexis Scale (BCS)" and "BETTER Model". Counselling programme of the women in the intervention group is held in four sessions one week apart and these women are provided with a counselling booklet accompanied by a CD. The scales are re-applied one month after the last session. In the control group, the women are left under routine hospital control after the scales are applied. The scales are re-applied to the control group after one month.

ELIGIBILITY:
Inclusion Criteria:

* who have had primary diagnosis of breast cancer and are at stage 0-I-II,
* who underwent mastectomy,
* who are in full remission, receiving no other treatment except hormonal therapy,
* who has been receiving hormonal treatment for at least two months and less than 5 years,
* age limit is set range from 18 to 45
* who are literate and sexually active,
* whose spouses had no sexual health problems,
* who don't have psychiatric illness
* who are capable of verbal communication and willing to participate in the study

Exclusion Criteria:

* who have had other cancer types or at stage III-IV
* who underwent conservative breast surgery
* who receive other treatment such as chemotherapy, radiotherapy
* above 45 years old
* who did not have sexual intercourse within the last month
* whose spouses have sexual health problems
* who have psychiatric illness
* who are not willing to participate in the study
* whose contact information could not be accessed

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
"Female Sexual Function Index" | 1.5 months
  "Female Sexual Function Index" has six subscales named as desire, arousal, lubrication, orgasm, satisfaction and pain. In subscales, increasing points evaluate positively. Scores between two and thirty-six are obtained from the scale. It is found to be a valid and reliable scale. "Female Sexual Function Index" scores of breast cancer patients who receive nursing counselling for sexual problems increase after counselling programme.
the functional scale of the "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast 23" | 1.5 months
  "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast 23" consists of 23 questions that look into the side effects of breast cancer treatments, body image, sexuality and future expectations. Scores between zero and one hundred points could be obtained from the scale. In Functional Scale increasing points evaluate positively. It is found to be a valid and reliable scale. The functional scale scores of the"European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast 23" of breast cancer patients who receive nursing counselling for sexual problems increase after counselling programme.
"Body Cathexis Scale" | 1.5 months
  This 40-item scale aims to measure the degree of happiness among people regarding their body sections and functions. Scores between 40 and 200 points can be obtained from the scale. This scale has no cut-off point. The high scores received indicate a high degree of satisfaction. Validity and reliability study for this scale is conducted in our country. "Body Cathexis Scale" scores of breast cancer patients who receive nursing counselling for sexual problems increase after counselling programme.
"Center for Epidemiologic Studies Depression Scale" | 1.5 months
  The scale consists of 20 items and four subscales on depression-related symptoms during a one week period. The total score that can be received from the scale vary between 0 and 60, with 16 points and above suggesting the probability of depression.It is a valid and reliable scale that is frequently used in cancer patients. "Center for Epidemiologic Studies Depression Scale" scores of breast cancer patients who receive nursing counselling for sexual problems decrease after the counselling programme.
The symptom scale of the "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast 23" | 1.5 months
  "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast 23" consists 23 questions that look into the side effects of breast cancer treatments, body image, sexuality and future expectations. Scores between zero and one hundred points could be obtained from the scale. In the Symptom Scales/Items decreasing points evaluate positively. It is found to be a valid and reliable scale. The symptom scale scores of the "European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast 23" of breast cancer patients who receive nursing counselling for sexual problems decrease after the counselling programme.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Olcer, Principal Investigator — Istanbul University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demirci S, Eser E, Ozsaran Z, Tankisi D, Aras AB, Ozaydemir G, Anacak Y. Validation of the Turkish versions of EORTC QLQ-C30 and BR23 modules in breast cancer patients. Asian Pac J Cancer Prev. 2011;12(5):1283-7. PMID 21875283
- [Result] Kedde H, van de Wiel HB, Weijmar Schultz WC, Wijsen C. Sexual dysfunction in young women with breast cancer. Support Care Cancer. 2013 Jan;21(1):271-80. doi: 10.1007/s00520-012-1521-9. Epub 2012 Jun 20. PMID 22714701
- [Result] Pinto AC. Sexuality and breast cancer: prime time for young patients. J Thorac Dis. 2013 Jun;5 Suppl 1(Suppl 1):S81-6. doi: 10.3978/j.issn.2072-1439.2013.05.23. PMID 23819031
- [Result] Krebber AM, Buffart LM, Kleijn G, Riepma IC, de Bree R, Leemans CR, Becker A, Brug J, van Straten A, Cuijpers P, Verdonck-de Leeuw IM. Prevalence of depression in cancer patients: a meta-analysis of diagnostic interviews and self-report instruments. Psychooncology. 2014 Feb;23(2):121-30. doi: 10.1002/pon.3409. Epub 2013 Sep 16. PMID 24105788
- [Result] Boquiren VM, Esplen MJ, Wong J, Toner B, Warner E, Malik N. Sexual functioning in breast cancer survivors experiencing body image disturbance. Psychooncology. 2016 Jan;25(1):66-76. doi: 10.1002/pon.3819. Epub 2015 Apr 27. PMID 25916689
- [Result] Mick J, Hughes M, Cohen MZ. Using the BETTER Model to assess sexuality. Clin J Oncol Nurs. 2004 Feb;8(1):84-6. doi: 10.1188/04.CJON.84-86. No abstract available. PMID 15043034
- [Result] Biglia N, Moggio G, Peano E, Sgandurra P, Ponzone R, Nappi RE, Sismondi P. Effects of surgical and adjuvant therapies for breast cancer on sexuality, cognitive functions, and body weight. J Sex Med. 2010 May;7(5):1891-900. doi: 10.1111/j.1743-6109.2010.01725.x. Epub 2010 Mar 2. PMID 20233281
- [Result] Panjari M, Bell RJ, Davis SR. Sexual function after breast cancer. J Sex Med. 2011 Jan;8(1):294-302. doi: 10.1111/j.1743-6109.2010.02034.x. Epub 2010 Sep 23. PMID 21199377
- [Result] Jun EY, Kim S, Chang SB, Oh K, Kang HS, Kang SS. The effect of a sexual life reframing program on marital intimacy, body image, and sexual function among breast cancer survivors. Cancer Nurs. 2011 Mar-Apr;34(2):142-9. doi: 10.1097/NCC.0b013e3181f1ab7a. PMID 20885305
- [Result] Perz J, Ussher JM; Australian Cancer and Sexuality Study Team. A randomized trial of a minimal intervention for sexual concerns after cancer: a comparison of self-help and professionally delivered modalities. BMC Cancer. 2015 Sep 9;15:629. doi: 10.1186/s12885-015-1638-6. PMID 26353787
- [Result] Rush CL, Darling M, Elliott MG, Febus-Sampayo I, Kuo C, Munoz J, Duron Y, Torres M, Galvan CC, Gonzalez F, Caicedo L, Napoles A, Jensen RE, Anderson E, Graves KD. Engaging Latina cancer survivors, their caregivers, and community partners in a randomized controlled trial: Nueva Vida intervention. Qual Life Res. 2015 May;24(5):1107-18. doi: 10.1007/s11136-014-0847-9. Epub 2014 Nov 8. PMID 25377349
- [Result] Kim GM, Kim SJ, Song SK, Kim HR, Kang BD, Noh SH, Chung HC, Kim KR, Rha SY. Prevalence and prognostic implications of psychological distress in patients with gastric cancer. BMC Cancer. 2017 Apr 20;17(1):283. doi: 10.1186/s12885-017-3260-2. PMID 28427439